CLINICAL TRIAL: NCT05462548
Title: The Safety and Efficiency of Luspatercept in Chinese Adults With Transfusion Dependent β-thalassemia: a Real-world Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianpei FANG, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-088-02
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Thalassemia Major; Transfusion-dependent Anemia
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Intervention Model Description: 18 years old or above
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- treatment group (Experimental): accept Luspatercept treatment
  Interventions: Drug: Luspatercept Injectable Product

INTERVENTIONS:
Drug: Luspatercept Injectable Product — 1-1.25mg/kg every 3 weeks subcutaneous injection
  Other Names: luspatercept

SUMMARY:
This is a prospective, single-arm, open-label study. Twenty adult patients with transfusion-dependent β -thalassemia will be enrolled to receive Luspatercept with optimal supportive care, including blood transfusion and iron removal, based on the clinician's judgment and practice. The main objective of this study was to evaluate the efficacy and safety of Luspatercept in the treatment of adult patients with transfusion-dependent β -thalassaemia in Chinese clinical practice, and to provide evidence reference for subsequent clinical use.

DETAILED DESCRIPTION:
Twenty adult patients with transfusion-dependent β -thalassemia will be enrolled to receive Luspatercept with optimal supportive care, being injected subcutaneously every 3 weeks ,by the dose of 1-1.25 mg/kg. The main objective of this study was to evaluate the efficacy and safety of Luspatercept in the treatment of adult patients with transfusion-dependent β -thalassaemia in Chinese clinical practice, and to provide evidence reference for subsequent clinical use.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years old

* The patient was clearly diagnosed as transfusion-dependent β -thalassemia, the blood transfusion period was ≤60 days, and the red blood cell infusion volume was not less than 3-12U in the 12 weeks before enrollment, which could provide the red blood cell infusion volume record in the 12 weeks before enrollment
* Patients who were treated with thalidomide before enrollment were required to stop the treatment for more than 4 weeks, and their hemoglobin decreased to below 90g/L. Blood transfusion was required, and records of blood transfusion within 12 weeks could be provided
* Voluntarily participate in the study and sign the informed consent;

Exclusion Criteria:

* (1) Pregnant or lactating women
* persons known to be allergic to Luspatercept and/or Luspatercept excipients for injection
* Severe liver dysfunction (liver enzyme (ALT or AST) ≥3 TIMES ULN)
* Severe renal impairment (eGFR < 30 ml/min/1.73m3 or patients with end-stage renal disease)
* Heart disease, heart failure classified as Class 3 or higher by the New York Heart Association (NYHA), or severe arrhythmia requiring treatment, or recent myocardial infarction within 6 months of randomization.
* The patient has uncontrolled hypertension. According to NCI CTCAE version 5.0, controlled hypertension in this protocol is considered to be ≤1.
* Patients with a history of deep vein thrombosis or stroke within 24 weeks prior to enrollment
* Erythropoietin, Luspatercept or hydroxyurea were used 8 weeks before enrollment
* Any other significant medical condition, laboratory abnormality, or mental illness that the Investigator deems inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
A 33% reduction in the red cell (RBC) transfusion burden for any 12 consecutive weeks within 24 weeks of Luspatercept treatment compared with baseline | 24 weeks
  the incidence of 33% reduction in RBC transfusion
The incidence of adverse events within 24 consecutive weeks of Luspatercept treatment | 24weeks
  incidence of reported adverse events

SECONDARY OUTCOMES:
the incidence of 50% reduction in transfusion in any 12 consecutive weeks | 24 weeks
  the incidence of 50% reduction in transfusion
Changes in mean cumulative transfusion volume from baseline at weeks 1-9, 1-12, and 1-24 | 24 weeks
  volume of transfusion
The rate of transfusion free at any 8 and 12 consecutive weeks in the entire study population | 24 weeks
  volume of transfusion
Changes in mean serum ferritin (SF) levels in the population from baseline | 24 weeks
  serum ferritin (SF) levels
Changes of cardiac and liver iron concentrations at 24 weeks from baseline (MRI T2*) | 24 weeks
  MR T2*
changes in reticulocyte levels from baseline during treatment | 24 weeks
  blood routine
changes in fetal hemoglobin levels from baseline during treatment | 24weeks
  Hemoglobin electrophoresis

CONTACTS AND LOCATIONS:
Overall Officials: Jianpei Fang, Dr., Study Director — SunYat-senU2H
Locations (1):
- The second affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
privacy information of individual participant is not available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: end of the study to 2 years after the end of study